CLINICAL TRIAL: NCT00750477
Title: A Multi-Center, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Effectiveness and Safety of Natural Eggshell Membrane (NEM) in the Treatment of Pain & Stiffness Associated With Moderate Osteoarthritis of the Knee
Brief Title: Efficacy & Safety Study Evaluating Natural Eggshell Membrane (NEM) in the Treatment of Osteoarthritis
Acronym: OPTION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ESM Technologies, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: CLN # C0504
Record Dates: First submitted 2008-09-08; First posted 2008-09-10 (Estimated); Last update posted 2016-02-15 (Estimated); Status verified 2016-02

CONDITIONS: Osteoarthritis
Keywords: osteoarthritis; arthritis; knee; eggshell; membrane; OPTION
MeSH Terms: conditions — Osteoarthritis; Arthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- NEM Treatment (Experimental): NEM, 500 mg, once daily, orally for 8 weeks
  Interventions: Dietary Supplement: NEM
- Placebo (Placebo Comparator): Placebo, 500 mg, once daily, orally for 8 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: NEM — see Treatment Arms
  Other Names: Natural Eggshell Membrane
  Arms: NEM Treatment
Dietary Supplement: Placebo — Placebo comparator containing inactives
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effectiveness of Natural Eggshell Membrane (NEM) for the relief of pain and stiffness associated with moderate osteoarthritis of the knee and to compare the effectiveness of NEM to placebo.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is the most prevalent form of arthritis and is estimated to affect nearly 27 million adults in the U.S., with one third of those 65 and older having been diagnosed with OA. As the population ages, this estimate is expected to grow rapidly. Traditional treatments for OA primarily attempt to address the symptoms (pain, inflammation, and discomfort) associated with the disease. This usually involves the use of analgesics (i.e. acetaminophen, tramadol), non-steroidal anti-inflammatory drugs (NSAIDs) (i.e. ibuprofen, diclofenac), or cyclooxygenase-2-specific (COX-2) NSAIDs (i.e. celecoxib) alone or in combination. Steroid and hyaluronic acid injections have also been used with some success. Many of these treatments have shown limited effectiveness in randomized controlled clinical trials (RCTs). To avoid the cardiac risks and gastrointestinal issues associated with traditional OA treatments (particularly with long-term use), many patients have turned to complementary and alternative medicines (CAMs) such as dietary supplements.

The discovery of eggshell membrane as a natural source of combined glucosamine, chondroitin, and hyaluronic acid has prompted the evaluation of this material as a potential treatment for OA. ESM Technologies, LLC (Carthage, MO) has developed methods to efficiently and effectively separate eggshell membrane from eggshells to create a shell-free eggshell membrane. The isolated membrane is then partially hydrolyzed using a proprietary process and dry-blended to produce 100% pure Natural Eggshell Membrane (NEM®).

In preliminary open-label human clinical trials totaling 37 subjects with OA, oral supplementation with 500 mg per day of NEM® resulted in an observed decrease in pain in 7-30 days. Therefore, an eight week randomized, multicenter, double blind, placebo controlled supplementation trial was conducted to evaluate the efficacy and safety of NEM® for the relief of the pain and stiffness associated with moderate OA of the knee - the Osteoarthritis Pain Treatment IncorpOrating NEM® (OPTION) trial.

ELIGIBILITY:
Inclusion Criteria:

* known symptomatic osteoarthritis of the knee
* patients must have been diagnosed with functional Grades I-III of osteoarthritis according to the modified criteria of the American College of Rheumatology
* must also have had persistent knee pain associated with osteoarthritis with a baseline score of at least 30 mm on the Patient's Assessment of Arthritis Pain - Visual Analog Scale
* required to suspend all current pain relief medications. Subjects that were currently taking analgesic medications were eligible to participate in the study following a 14 day washout period for NSAIDs, a 7 day washout for narcotics, and a 90 day washout for injected steroids. Subjects currently taking glucosamine, chondroitin sulfate or MSM were only eligible after a 3-month washout period.

Exclusion Criteria:

* are currently receiving remission-inducing drugs such as methotrexate or immunosuppressive medications or had received them within the past 3 months
* had a confounding inflammatory disease or condition (rheumatoid arthritis, gout, pseudo gout, Paget's disease, chronic pain syndrome, etc.) that would interfere with assessment of pain associated with the index knee
* body weight 250 pounds or greater
* having a known allergy to eggs or egg products
* pregnant or breastfeeding women
* Subjects previously enrolled in a study to evaluate pain relief within the past 6 months or currently involved in any other research study involving an investigational product (drug, device, or biologic) or a new application of an approved product, within 30 days of screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2004-12; Primary Completion 2006-01 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of the study was measurement of the effectiveness of NEM® in relieving pain, stiffness, and discomfort associated with moderate OA of the knee and to compare its effectiveness to placebo. | 10, 30, & 60 Days

SECONDARY OUTCOMES:
Secondary objectives of the study were to evaluate tolerability and any adverse reactions associated with supplementation with NEM®. | 10, 30, & 60 Days

CONTACTS AND LOCATIONS:
Overall Officials: Anne Winkler, MD, PhD, Principal Investigator — St. John's Clinic - Rheumatology; Robert W Jackson, DO, Principal Investigator — Regional Specialty Clinic; Kevin J Ruff, PhD, MBA, Study Director — ESM Technologies, LLC
Locations (3):
- United States (3):
  - Regional Specialty Clinic, Cuba, Missouri
  - Regional Specialty Clinic, Kirksville, Missouri
  - St. John's Clinic, Springfield, Missouri

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ruff KJ, Winkler A, Jackson RW, DeVore DP, Ritz BW. Eggshell membrane in the treatment of pain and stiffness from osteoarthritis of the knee: a randomized, multicenter, double-blind, placebo-controlled clinical study. Clin Rheumatol. 2009 Aug;28(8):907-14. doi: 10.1007/s10067-009-1173-4. Epub 2009 Apr 2. PMID 19340512
- See also: Digital Object Identifier link to published study in Clinical Rheumatology. — http://dx.doi.org/10.1007/s10067-009-1173-4